CLINICAL TRIAL: NCT07058168
Title: The Effect of Labor Diet Administered to Multiparous Pregnant Women on Mother and Baby During the Delivery Process
Brief Title: The Effect of Labor Diet During the Delivery Process
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Nilgun Avci, Biruni Unşversity, Biruni University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-KAEK-54-21-06
Record Dates: First submitted 2025-06-13; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Labor Pain; Labor; Diet
Keywords: labor; diet; labor diet; pregnant; delivery
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: The study population consisted of all multiparous pregnant women admitted to the maternity unit of a state hospital on the European side of Istanbul between February and June 2022. Power analysis (G*Power 3.1 program) was used to determine the sample. As a result of the analysis (with an effect size of 0.932, a confidence interval of 95%, and an error of 0.05), it was found that at least 47 pregnant women should be included in a group (12). Ninety-four pregnant women (experimental group:47; control group:47) were included in the sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: This research is planned with experimental design (Experimental): The data collection tools "Personal Information Form", "Women's Perception of Supportive Care Provided at Birth Scale", and "Pregnant and Infant Monitoring Form (VAS pain, anxiety, fatigue and thirst scales)" were applied. The VAS scales contains numbers evenly spaced (0-10) on a line. It's an evaluation scale filled out by pregnants stating their current levels by givig a number. The cut off point of the VAS anxiety and thirst scales were found to be four.In VAS anxiety, scores above this cut-off point indicate deviation from normal and individuals must be handled by professionals. In VAS thirst, patients who score above this score are considered to be experiencing dehydration symptoms. The time of the last meal was learnt according to the information given by the pregnant woman. Spontaneous blood glucose measurement was performed in all pregnant women. Intermittent NST follow-up and routine medical treatment were continued.
  Interventions: Dietary Supplement: Other: experimental group (labor diet)

INTERVENTIONS:
Dietary Supplement: Other: experimental group (labor diet) — The data collection tools "Personal Information Form", "Women's Perception of Supportive Care Provided at Birth Scale", and "Pregnant and Infant Monitoring Form (VAS pain, anxiety, fatigue and thirst scales)" were applied. The VAS scales contains numbers evenly spaced (0-10) on a line. It's an evaluation scale filled out by pregnants stating their current levels by givig a number. The cut off point of the VAS anxiety and thirst scales were found to be four.In VAS anxiety, scores above this cut-off point indicate deviation from normal and individuals must be handled by professionals. In VAS thirst, patients who score above this score are considered to be experiencing dehydration symptoms. The time of the last meal was learnt according to the information given by the pregnant woman. Spontaneous blood glucose measurement was performed. The labor diet was administered after 6 hours of fasting. Post-prandial blood glucose and tools were measured after the labor diet (at the 2nd hours)

SUMMARY:
This study is a clinical trial. It aimed to examine the effects of the labor diet on pain, anxiety, fatigue, and thirst levels, maternal satisfaction during labor, in multiparous pregnant women (47 experiments; 47 controls) in the first stage of labor. Criteria for inclusion in the study: Pregnant women with cervical dilatation less than 5 cm, and who were suitable for oral intake, and voluntarily accept to participate in the research were included in the study. Exclusion criteria from the study: Exclusion criteria from the study: Pregnant women who have auditory or mental health problems; who could not speak or understand Turkish, who were under 18 years of age, who were primiparous, who were chronically ill and whose current pregnancy was risky. The pain, anxiety, fatigue, and thirst levels of the pregnant women in the control group were evaluated with scales every two hours during labour. Pregnant women in the experimental group labor diet and their pain, anxiety, fatigue and thirst levels were evaluated with scales every two hours until labor. The main questions it aims to answer are: • Labor diet during labor; It is effective in reducing the level of pain. • Labor diet during labor; It is effective in reducing anxiety. • Labor diet during labor; It is effective in reducing thirst. • Labor diet during labor; It is effective in reducing fatigue. • Labor diet during labor; It is effective in increasing maternal satisfaction. Routine medical treatment of pregnant women continued all groups. Only pregnant women who in the experimental group labor diet also.

DETAILED DESCRIPTION:
Objective: In this study, it was aimed to examine the effects of the labor diet on pain, anxiety, fatigue, and thirst levels, maternal satisfaction during labor, in multiparous pregnant women in the first stage of labor. Methods: The study was conducted in a randomized controlled experimental manner. The universe consisted of all pregnant women who applied to the delivery room of a public institution between February and June 2022. Power analysis was used to determine the sample. 94 pregnant women (47 experiments;47 controls) were included in the study. The study was started after the approval of the ethics committee and the institution. As a data collection tool in the research; "Personal Information Form","Women's Perception of Supportive Care Provided at Birth Scale" and "Pregnant and Infant Monitoring Form" were used.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal delivery,
* Who volunteered to participate in the research,
* Who with cervical dilatation less than 5 cm,
* who were suitable for oral intake

Exclusion Criteria:

* Who could not speak or understand Turkish,
* Have auditory or mental health problems,
* Who were under 18 years of age,
* Who were primiparous,
* Who were chronically ill and whose current pregnancy was risky

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Anxiety VAS (vizual scale) | Time Frame: Anxiety scale used starting to labor diet. The delivery diet was administered according to the completion of the 6-hour fasting period. At 2 hours after the diet intake, the scale was repeated.
  Description: Change from anxiety scale scores at control group or experimental group in during labor. The minimum score is 0 and the maximum score is 10. The higher the score, the greater the person's anxiety.
Fatigue VAS (vizual scale) | Time Frame: Fatigue scale used starting to labor diet. The delivery diet was administered according to the completion of the 6-hour fasting period. At 2 hours after the diet intake, the scale was repeated.
  Description: Change from fatigue scale scores at control group or experimental group in during labor. The minimum score is 0 and the maximum score is 10. The higher the score, the greater the person's fatigue.

SECONDARY OUTCOMES:
Pain VAS (Vizual scale) | Time Frame: Pain scale used starting to labor diet. The delivery diet was administered according to the completion of the 6-hour fasting period. At 2 hours after the diet intake, the scale was repeated.
  Description: Change from pain scale scores at control group or experimental group in during labor. The minimum score is 0 and the maximum score is 10. The higher the score, the greater the person's pain.
Thirst VAS (Vizual scale) | Time Frame: Thirst scale used starting to labor diet. The delivery diet was administered according to the completion of the 6-hour fasting period. At 2 hours after the diet intake, the scale was repeated.
  Description: Change from thirst scale scores at control group or experimental group in during labor. The minimum score is 0 and the maximum score is 10. The higher the score, the greater the person's thirst.

CONTACTS AND LOCATIONS:
Overall Officials: nilgün avcı, Principal Investigator — Biruni University
Locations (1):
- Biruni University, Zeytinburnu, Istanbul, Turkey (Türkiye)